CLINICAL TRIAL: NCT03168191
Title: Flavors and E-cigarette Effects in Adolescent Smokers- STUDY 2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 1307012312-2
Record Dates: First submitted 2017-04-27; First posted 2017-05-30 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine; Menthol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- E-cigarette flavor (Experimental): In this arm, subjects will receive an experimental flavor. Participants will be randomly assigned to low or high dose of nicotine.
  Interventions: Drug: Nicotine; Other: Experimental Flavor
- Menthol Flavor (Experimental): In this arm, subjects will receive a menthol flavor. Participants will be randomly assigned to low or high dose of nicotine.
  Interventions: Drug: Nicotine; Other: Menthol Flavor
- No Flavor (Placebo Comparator): In this arm, subjects will receive no flavor. Participants will be randomly assigned to low or high dose of nicotine.
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Nicotine — Participants will receive low dose nicotine (6 mg/ml) or high dose nicotine (12 mg/ml)
Other: Experimental Flavor — Experimental fruit flavored e-cigarette for lab session
  Arms: E-cigarette flavor
Other: Menthol Flavor — Menthol flavored e-cigarette for lab session
  Arms: Menthol Flavor

SUMMARY:
This study is to examine if inhaled doses of an e-cigarette flavor, alone and in combination with menthol, changes the appeal of e-cigarettes containing low and high doses of nicotine. The hypothesis is that menthol and the other experimental flavor will interact with nicotine dose to improve taste and liking for e-cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-20 years
* Able to read and write
* Urine cotinine levels of >250 ng/ml at screening appointment
* Use of e-cigarettes in the past month
* May or may not currently smoke traditional cigarettes

Exclusion Criteria:

* Seeking smoking cessation treatment
* Current/lifetime criteria for dependence on another psychoactive substance -Daily use of alcohol or marijuana or use of any other drugs including cocaine, opiates, stimulants
* Regular use of psychoactive drugs including anxiolytics, antidepressants and other psychostimulants
* Current or past history of psychosis or other psychiatric diagnosis such as major depression
* Any significant current medical condition

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Change score in Liking/wanting of the e-cigarette | Baseline (+10 minutes) to end of lab session (+40 minutes)
  The Drug Effects Questionnaire (Soria et al) will be used to ask about liking and wanting during the lab session

SECONDARY OUTCOMES:
Change score in rating of coolness | Baseline (+10 minutes) to end of lab session (+40 minutes)
  gMLS rating of e-cigarette coolness
Change score in rating of harshness/irritation | Baseline (+10 minutes) to end of lab session (+40 minutes)
  gMLS rating of e-cigarette harshness/irritation
Change score in rating of sweetness | Baseline (+10 minutes) to end of lab session (+40 minutes)
  gMLS rating of e-cigarette sweetness
Change score in rating of sourness | End of lab session (+40 minutes)
  gMLS rating of e-cigarette sourness
Change score in rating of fruitiness | Baseline (+10 minutes) to end of lab session (+40 minutes)
  gMLS rating of e-cigarette fruitiness
Change score in rating of total sensation | Baseline (+10 minutes) to end of lab session (+40 minutes)
  gMLS rating of e-cigarette total sensation
E-cigarette value | Baseline (+10 minutes) to end of lab session (+40 minutes)
  Value of e-cigarette as determined by the Multiple Choice Questionnaire (MCP) task
Number of puffs | End of ad-lib lab session 4 (+40 minutes)
  Number of puffs taken at the end of the ad-lib vaping period
Change score in Tobacco Craving | Baseline (+10 minutes) to end of lab session (+40 minutes)
  The Brief Questionnaire on Smoking Urges (Tiffany & Drobes,1991) will be used to assess the magnitude of change in tobacco craving during the lab session

CONTACTS AND LOCATIONS:
Overall Officials: Dana Cavallo, Ph.D., Study Director — Yale University
Locations (1):
- CMHC, Substance Abuse Center, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Jackson A, Green B, Erythropel HC, Kong G, Cavallo DA, Eid T, Gueorguieva R, Buta E, O'Malley SS, Krishnan-Sarin S. Influence of menthol and green apple e-liquids containing different nicotine concentrations among youth e-cigarette users. Exp Clin Psychopharmacol. 2021 Aug;29(4):355-365. doi: 10.1037/pha0000368. Epub 2020 Apr 16. PMID 32297782